CLINICAL TRIAL: NCT06707571
Title: Ultrasongraphy Guided Spinal Anesthesia Versus Landmark in Lower Abdominal Surgeries in Cancer Patients: a Randomized Controlled Trial
Brief Title: Landmark Versus Ultrasongraphy Guided Spinal Anesthesia in Lower Abdominal Surgeries in Cancer Patients: a Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maram Ashraf Zahr Eldeen, Anesthesia, Intensive Care and Pain Management Department South Egypt cancer Institute, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: landmark VS US guided
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Cancer Surgery
Keywords: US-guided spinal anesthesia
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be randomly assigned to receive spinal anesthesia using the surface landmark-guided (landmark group) or preprocedural ultrasound-assisted (ultrasound group) technique using a computer-generated table of random numbers. Group allocation will be concealed by sequentially numbered, sealed opaque envelopes, which are opened only by the attending anesthesiologist immediately before the procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Landmark Group (Experimental): patients will receive spinal anesthesia using the surface landmark-guided
  Interventions: Procedure: spinal anesthesia
- Ultrasonography Group (Experimental): patients will receive spinal anesthesia after us-assisted technique
  Interventions: Procedure: spinal anesthesia

INTERVENTIONS:
Procedure: spinal anesthesia — spinal anesthesia after us-assisted technique
  Arms: Ultrasonography Group
Procedure: spinal anesthesia — spinal anesthesia using the surface landmark-guided
  Arms: Landmark Group

SUMMARY:
Spinal anesthesia is a commonly employed technique for lower abdominal surgeries, providing effective anesthesia and analgesia with minimal systemic effects. In cancer patients undergoing such procedures, careful consideration of anesthetic techniques is crucial, given their often-compromised physiological state and the need to minimize postoperative complications. Two approaches to administering spinal anesthesia are Ultrasound (US)-guided and the traditional landmark-based technique.

the aim of the study :To evaluate the efficacy, safety and feasibility of US-guided spinal anesthesia versus the landmark-based technique in cancer patients undergoing lower abdominal surgery.

DETAILED DESCRIPTION:
The traditional landmark method relies on palpating anatomical structures, such as the iliac crests and spinal processes, to guide needle insertion. Although widely used, it can be challenging in patients with anatomical variations, obesity, or previous surgeries, potentially leading to multiple attempts, increased patient discomfort, or complications. On the other hand, Ultrasound (US) imaging has become an increasingly popular tool among anesthesiologists to guide neuraxial blockade. US-guided spinal anesthesia provides real-time visualization of the relevant anatomy, including the spinal canal, ligaments, and surrounding tissues, enabling more accurate needle placement. This technique has gained attention for its potential to improve success rates, reduce complications, and enhance patient comfort, particularly in complex cases such as cancer patients, where precision is vital.

By examining factors such as procedural success rates, patient comfort, complication rates, and overall outcomes, we can better understand the role of ultrasound guidance in optimizing anesthetic care for this vulnerable patient population.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Both sex
* patients with a body mass index (BMI) of 18-40 kg/m2
* American Society of Anesthesiologists (ASA) physical status classification of I to III.

Exclusion Criteria:

* • Patients have a contraindication for regional anesthesia, e.g. coagulopathy.

  * Failed or unsatisfactory intrathecal block.
  * Patients with known hypersensitivity to amide local anesthetics.
  * Local injection site infection or spinal deformity.
  * Severe hypotension.
  * Space occupying lesions of the brain.
  * Hypovolemia.
  * Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
the first-pass success rate of Combined spinal-epidural anesthesia | baseline
  first-pass success was defined as the needle reaching the subarachnoid space within a single insertion attempt, without redirection

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Park SK, Yoo S, Kim WH, Lim YJ, Bahk JH, Kim JT. Ultrasound-assisted vs. landmark-guided paramedian spinal anaesthesia in the elderly: A randomised controlled trial. Eur J Anaesthesiol. 2019 Oct;36(10):763-771. doi: 10.1097/EJA.0000000000001029. PMID 31188153
- [Background] Li M, Ni X, Xu Z, Shen F, Song Y, Li Q, Liu Z. Ultrasound-Assisted Technology Versus the Conventional Landmark Location Method in Spinal Anesthesia for Cesarean Delivery in Obese Parturients: A Randomized Controlled Trial. Anesth Analg. 2019 Jul;129(1):155-161. doi: 10.1213/ANE.0000000000003795. PMID 30234528
- [Background] Coviello A, Iacovazzo C, Piccione I, Posillipo C, Barone MS, Ianniello M, de Siena AU, Cirillo D, Vargas M. Impact of Ultrasound-Assisted Method on Success Rate of Spinal Anesthesia Performed by Novice Trainees: A Retrospective Comparative Study. J Pers Med. 2023 Oct 21;13(10):1515. doi: 10.3390/jpm13101515. PMID 37888126
- [Background] Geng J, Chen XL, Wang XD, Guo XY, Li M. [Ultrasound imaging increases first-attempt success rate of neuraxial block in elderly patients]. Zhonghua Yi Xue Za Zhi. 2016 Nov 22;96(43):3459-3463. doi: 10.3760/cma.j.issn.0376-2491.2016.43.004. Chinese. PMID 27903338
- [Background] Zhu G, Wang X, Yang L. Real-time ultrasound-guided neuraxial anesthesia for cesarean section in parturients with previous internal fixation surgery for lumbar fracture: a case series. Quant Imaging Med Surg. 2023 Jan 1;13(1):529-535. doi: 10.21037/qims-22-223. Epub 2022 Oct 26. No abstract available. PMID 36620151
- [Background] Sahin T, Balaban O, Sahin L, Solak M, Toker K. A randomized controlled trial of preinsertion ultrasound guidance for spinal anaesthesia in pregnancy: outcomes among obese and lean parturients: ultrasound for spinal anesthesia in pregnancy. J Anesth. 2014 Jun;28(3):413-9. doi: 10.1007/s00540-013-1726-1. Epub 2013 Oct 20. PMID 24141882
- [Background] Feng Q, Zhang L, Zhang M, Wen Y, Zhang P, Wang Y, Zeng Y, Wang J. Morphological parameters of fourth lumbar spinous process palpation: a three-dimensional reconstruction of computed tomography. J Orthop Surg Res. 2020 Jun 22;15(1):227. doi: 10.1186/s13018-020-01750-2. PMID 32571368